CLINICAL TRIAL: NCT02548559
Title: Sublingual Cannabidiol for Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Staci Gruber, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Staci Gruber, Ph.D., Director, Cognitive and Clinical Neuroimaging Core, Mclean Hospital
Organization: Mclean Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P000959
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Full-Spectrum Cannabidiol (Experimental): 1 ml of full-spectrum sublingual cannabidiol solution (10 mg/ml CBD) administered three times per day (TID) for four weeks.
  Interventions: Drug: Full-Spectrum Cannabidiol
- Single-Compound Cannabidiol (Experimental): 1 ml of single-compound sublingual cannabidiol solution (10 mg/ml CBD) administered three times per day (TID) for four weeks.
  Interventions: Drug: Single-Compound Cannabidiol
- Placebo (Placebo Comparator): 1 ml of placebo solution administered three times per day (TID) for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Full-Spectrum Cannabidiol — Full-Spectrum Cannabidiol; total daily dose of 30 mg.
  Arms: Full-Spectrum Cannabidiol
Drug: Single-Compound Cannabidiol — Single-Compound Cannabidiol; total daily dose of 30 mg.
  Arms: Single-Compound Cannabidiol
Drug: Placebo — Placebo solution.
  Arms: Placebo

SUMMARY:
This is an open-label to double-blind study evaluating the effects of cannabidiol (CBD) for the treatment of anxiety in adults. Participants will use a sublingual (under-the-tongue) solution of whole plant-derived CBD or placebo three times daily for four weeks in addition to their normal treatment regimen. Participants' clinical state will be assessed weekly during the treatment period. In addition, cognitive function and measures of quality of life, sleep, and general health will be assessed at baseline and the post-treatment final visit.

DETAILED DESCRIPTION:
Cannabis has been used for medicinal purposes across many cultures for a range of disorders for thousands of years. The plant is comprised of a variety of components, such as phytocannabinoids, which include (among others) the major intoxicating constituent of cannabis, delta-9 tetrahydrocannabinol (THC), and cannabidiol (CBD), a major non-intoxicating constituent of cannabis. Increasing evidence indicates that CBD in particular may have significant medicinal properties and benefits; experimental studies in both animals and humans have demonstrated that CBD can act as an anticonvulsant, antipsychotic, and muscle relaxant. Several studies have demonstrated that CBD produces acute anxiolytic effects in animals and humans, although thus far no clinical trials of CBD have been conducted in patients with anxiety. As a growing number of states are legalizing medical cannabis, a gap exists in the scientific literature regarding the effects of CBD on anxiety.

This investigation is composed of two stages. Stage 1 is comprised of a four-week, open-label clinical trial of a high-CBD containing compound in individuals with anxiety. Participants will be pre-screened by phone in order to evaluate their eligibility for the study. If approved, participants will come to the hospital for a baseline/screening visit, and will complete a structured clinical interview, clinical and quality of life questionnaires, and cognitive assessments. Enrolled participants will be given CBD solution to use for the duration of the study; participants will be instructed to self-administer 1 milliliter (ml) of the tincture under the tongue three times per day for four weeks. Throughout the treatment period, participants will return to the hospital on a weekly basis to complete questionnaires about their mood and quality of life. Participants will also return to the hospital for a final visit after four weeks of treatment to complete additional questionnaires and cognitive assessments. Stage 1 of the study was completed in early 2020.

Stage 2 of the study is a double-blind clinical trial of this solution in patients with anxiety. This double-blind trial began after the open-label trial was completed. In the same manner as the open-label trial, participants will be pre-screened by phone, and approved participants will come to the hospital for a baseline/screening visit to complete a structured clinical interview, questionnaires, and cognitive assessments. Eligible participants will also have the option to complete an hour-long MRI scan at the baseline and final visits. Enrolled participants will receive either full-spectrum CBD solution, single-compound CBD solution, or placebo solution to self-administer throughout the four week treatment period, as described above. Participants will return to the hospital weekly during the treatment period to complete questionnaires about their mood and quality of life. Participants in this stage of the study will also return for a final visit after four weeks of treatment to complete additional questionnaires, cognitive assessments, and an optional hour-long MRI scan. We are currently recruiting for Stage 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Native English speaker or acquired English prior to age 5
* Provides informed consent
* Endorses moderate or severe anxiety at the screening visit

Exclusion Criteria:

* Non-native English speakers
* Estimated IQ < 75
* Pregnancy
* Presence of serious medical illness, including liver or kidney disease, neurological disorder, or certain psychiatric disorders
* History of head injury or loss of consciousness >5 minutes
* Current use of cannabis or cannabinoid products >1x/month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Reported Anxiety as Assessed by the Beck Anxiety Inventory (BAI) | Week 1, Week 2, Week 3, Week 4
  The BAI is a 21-item self-report measure used to rate subjective, somatic, and panic-related symptoms of anxiety on a scale of 0 to 3 (higher scores indicating more anxiety).
Change from Baseline in Anxiety Assessed by the Overall Anxiety Severity and Impairment Scale (OASIS) | Week 1, Week 2, Week 3, Week 4
  The OASIS is a brief 5-item measure used to evaluate the functional impairment cause by anxiety that will be given on a weekly basis; the frequency and intensity of anxiety, as well as the degree of avoidance and interference with work and social function are rated on a scale of 0 to 4 (higher scores indicating more anxiety).
Change from Baseline in Self-Reported Anxiety Assessed by the State-Trait Anxiety Inventory (STAI) | Week 1, Week 2, Week 3, Week 4
  This self-report measure is comprised of two 20-item scales, with a range of four possible responses from 1 to 4 (higher scores indicating more anxiety), and differentiates between the more temporary condition of "state" anxiety and the more general quality of "trait" anxiety.
Change from Baseline in Anxiety Measured by the Hamilton Anxiety Scale (HAM-A) | Week 1, Week 2, Week 3, Week 4
  This observer-rating 14-item scale is administered in the form of an interview, and allows information from multiple sources to influence ratings (i.e. subject report, examiner's observation), and has been shown to be reliable index of clinical state. A range of 5 possible responses (0-4, not present-very severe) are possible for each item.

SECONDARY OUTCOMES:
Change from Baseline in Depressive Symptoms Assessed by the Beck Depression Inventory (BDI) | Week 1, Week 2, Week 3, Week 4
  The BDI is a 21 item-self-report measure that can be used to assess the severity of depression. Each item on the BDI relates to a symptom of depression and is rated by the subject using a 0-3 scale (higher scores indicating increased severity).
Change from Baseline in Sleep Quality Assessed by the Pittsburgh Sleep Quality Index (PSQI) | Week 1, Week 4
  The PSQI contains 19 self-rated questions that assess sleep quality and disturbance over the previous 1-month period. The 19 items yield seven component scores such as sleep latency, sleep duration, and daytime dysfunction, which are then summed to generate a global score (higher scores indicating decreased sleep quality).
Change from Baseline in Mood Measured by the Profile of Mood States (POMS) | Week 1, Week 2, Week 3, Week 4
  Comprised of 72 adjectives commonly used to describe mood states, subjects are asked to indicate how they feel at that moment in relation to each of the adjectives using a five point scale ranging from "not at all" (0) to "extremely" (4). The POMS consists of 10 scales, which measure friendliness, anxiety, depression, fatigue, anger, elation, confusion, vigor, arousal, and positive mood.
Change from Baseline in Mood Assessed by the Positive and Negative Affect Scale (PANAS) | Week 1, Week 2, Week 3, Week 4
  The PANAS is a 20-item self-report scale in which mood variables are rated by subjects on a 1-5 scale (from very slightly/not at all to extremely), based on how they feel. Ten PANAS items rate positive affect (PA), that is, the extent to which a person feels enthusiastic, active, and alert; ten items rate negative affect (NA), that is, the extent to which a person is experiencing subjective distress and aversive mood states.
Change from Baseline in Quality of Life Measured by the 36-Item Short Form (SF-36) | Week 1, Week 4
  The SF-36 is a multi-purpose, 36-item short-form health survey that gives an 8-scale profile of functional health and well-being scores (higher scores indicate better quality of life).
Change from Baseline in Sexual Health Measured by the Arizona Sexual Experience Scale (ASEX) | Week 1, Week 4
  The ASEX contains 5 items designed to assess sexual health and sexual dysfunction. The scale contains both a male and female version, with only one question different. Each item is scored on a scale from 1-6, with higher scores indicating increased dysfunction.
Patient's Global Impression of Change (PGIC) Scale Score at Week 4 | Week 4
  The PGIC is a single-question, 7-point scale depicting a patient's rating of overall improvement from "very much worse" to "very much improved".
Change from Baseline on Stroop Color-Word Test | Week 1, Week 4
  This test measures the ability to inhibit inappropriate responses and resist interference. Increased errors and time to complete the test reflect poorer performance.
Change from Baseline on Trail Making Test | Week 1, Week 4
  This test is designed to measure visual conceptual and visuomotor tracking, as well as maintenance of cognitive set. Increased errors and time to complete the test reflect poorer performance.
Change from Baseline on the Wisconsin Card Sort Test (WCST) | Week 1, Week 4
  This test assesses a person's ability to form abstract concepts, utilize feedback, and to shift and maintain set. Total number of categories correct, perseverative and other error types are calculated, with increased errors and decreased number of categories correct indicating poorer performance.
Change from Baseline on the Multi-Source Interference Task (MSIT) | Week 1, Week 4
  This test assesses a person's ability to ignore distracting stimuli and identify the correct item. Increased numbers of errors indicate poorer performance.
Change from Baseline on the Letter-Number Sequencing (LNS) Subtest of the Wechsler Adult Intelligence Scale | Week 1, Week 4
  This subtest is designed to assess working memory and primarily measures the efficiency of attention, concentration and mental control. Higher scores reflect better performance.
Change from Baseline on the Digit Symbol Substitution Test (DSST) of the Wechsler Adult Intelligence Scale | Week 1, Week 4
  The DSST measures attention, psychomotor speed, visual scanning and information processing. Higher scores reflect better performance.
Change from Baseline on the Controlled Oral Word Association Test (COWAT) | Week 1, Week 4
  This test measures the subject's ability to produce individual words under restricted conditions, and interrogates both executive function and verbal memory. Performance is measured by an age and education corrected total of the number of words generated for each section, with higher numbers indicating better performance.
Change from Baseline on the Rey Auditory Verbal Learning Test (RAVLT) | Week 1, Week 4
  This verbal learning test assesses the subject's immediate and delayed recall. Higher scores reflect better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Staci Gruber, PhD., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital Brain Imaging Center, Belmont, Massachusetts, United States